CLINICAL TRIAL: NCT03512834
Title: Phase II Trial, Multicenter, First Line Paclitaxel-Avelumab Treatment for Inoperable Angiosarcoma
Brief Title: Paclitaxel-Avelumab for Angiosarcoma
Acronym: ASAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sung Yong Oh (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor-Investigator, Sung Yong Oh, Dong-A University Hospital, Dong-A University Hospital
Organization: Dong-A University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAUHIRB-18-052
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Angiosarcoma Metastatic
Keywords: angiosarcoma; paclitaxel; avelumab
MeSH Terms: conditions — Hemangiosarcoma | interventions — avelumab; Paclitaxel; genexol-PM

STUDY DESIGN:
Intervention Model Description: Paclitaxel + Avelumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paclitaxel+Avelumab (Experimental): Paclitaxel combination with Avelumab for inoperable angiosarcoma
  Interventions: Drug: Avelumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Avelumab — Avelumab 10mg/kg, administered via I.V infusion over 1hour, every 2weeks until disease progression or unacceptable toxicity
  Other Names: BAVENCIO
Drug: Paclitaxel — Paclitaxel 80mg/m2 D1,8 and 15 , administered via I.V infusion, every 4 weeks.
  Other Names: TAXOL; GENEXOL; ANZATAX

SUMMARY:
To investigate the efficacy of Avelumab when given in combination with paclitaxel as a first line treatment for the patients with inoperable angiosarcoma.

DETAILED DESCRIPTION:
Angiosarcomas are very rare tumors (incidence < 1/100.000/year) of vascular or lymphatic origin characterized by a clinical heterogeneity in terms of presentation and behavior.In several prospective and retrospective studies, weekly paclitaxel showed promising activity in patients with advanced or metastatic angiosarcoma. Given the important role of PD-L1 in the suppression of T-cell responses, and the mode of action of avelumab which blocks the interaction between PD-L1 and its receptors, avelumab is being developed as a potential therapy for subjects with various tumors. In prior study cutaneous angiosarcoma patients with a high infiltration of PD-1-positive cells with tumor site PD-L1 expression were more likely to have favorable survival.

Therefore, antitumor activity of Avelumab as inhibitor of PD-1/PDL-1 interaction with Paclitaxel, standard chemotherapy, might have more therapeutic improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Male or female subjects aged ≥ 20 years.
3. Histologically or cytologically proven metastatic or locally advanced Angiosarcoma.
4. Inoperable Angiosarcoma
5. Chemo-naïve patient
6. ECOG performance status of 0 to 1 at trial entry and an estimated life expectancy of at least 3 months.
7. Disease must be measurable with at least 1 measurable lesion by RECIST 1.1
8. Adequate hematological function defined by white blood cell (WBC) count ≥ 3 × 109/L with absolute neutrophil count (ANC) ≥ 1.5 × 109/L, lymphocyte count ≥ 0.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused).
9. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal range (ULN), an aspartate aminotransferase (AST), level ≤ 2.5 × ULN, and an alanine aminotransferase (ALT) level ≤ 2.5 × ULN or, for subjects with documented metastatic disease to the liver, AST and ALT levels

   ≤ 5 × ULN.
10. Adequate renal function defined by an estimated creatinine clearance > 30mL/min according to the Cockcroft-Gault formula.
11. Highly effective contraception (that is, methods with a failure rate of less than 1% per year) for both male and female subjects if the risk of conception exists

Exclusion Criteria:

1. Concurrent treatment with a non-permitted drug (see Section 14)
2. Prior therapy with any antibody/drug targeting T cell co-regulatory proteins (immune checkpoints) such as anti-PD-1, anti-PD-L1, or anti-cytotoxic T-lymphocyte antigen-4 (CTLA-4) antibody.
3. Concurrent anticancer treatment within 28 days before the start of trial treatment (e.g., cytoreductive therapy, radiotherapy [with the exception of palliative bone directed radiotherapy], immune therapy, or cytokine therapy except for erythropoietin)
4. Major surgery within 28 days before the start of trial treatment (excluding prior diagnostic biopsy)
5. Use of hormonal agents within 7 days before the start of trial treatment.
6. Use of any investigational drug within 28 days before the start of trial treatment.
7. Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of the study treatment (with the exception of patients with adrenal insufficiency, who may continue corticosteroids at physiologic replacement dose, equivalent to ≤ 10 mg prednisone daily). Steroids with no or minimal systemic effect (topical, inhalation) are allowed.
8. Previous malignant disease other than the target malignancy to be investigated in this trial within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ.
9. Rapidly progressive disease (e.g., tumor lysis syndrome).
10. Active or history of central nervous system (CNS) metastases.
11. Receipt of any organ transplantation including allogeneic stem-cell transplantation.
12. Significant acute or chronic infections including, among others:

    1. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
    2. Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive).
13. Active or history of any autoimmune disease (subjects with diabetes Type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible) or immunodeficiencies.
14. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI-CTCAE v4.0), any history of anaphylaxis, or uncontrolled asthma (i.e., 3 or more features of partly controlled asthma).
15. Persisting toxicity related to prior therapy Grade > 1 NCI-CTCAE v4.0, however sensory neuropathy

    ≤ Grade 2 is acceptable.
16. Pregnancy or breast feeding.
17. Known alcohol or drug abuse.
18. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication.
19. All other significant diseases (e.g., inflammatory bowel disease), which, in the opinion of the investigator, might impair the subject's tolerance of trial treatment.
20. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
21. Legal incapacity or limited legal capacity.
22. Vaccination within 4 weeks of the first dose of avelumab and while on study is prohibited except for administration of inactivated vaccines (e.g. inactivated influenza vaccines).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | up to 6 months
  CR+PR by RECIST

SECONDARY OUTCOMES:
Progression free survival | up to 12 months
  progression or death
Overall survival | up to 12 months
  death event
Adverse event | up to 12 months
  By NCI-CTC v4.03

CONTACTS AND LOCATIONS:
Overall Officials: SUNG YONG OH, MD, Principal Investigator — Dong-A University Hospital
Locations (1):
- Sung Yong Oh, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No